CLINICAL TRIAL: NCT01803425
Title: Post-marketing Surveillance (PMS) of GlaxoSmithKline Biologicals' 10-valent Pneumococcal Conjugate Vaccine (Synflorix™) When Administered to Healthy Infants and Children According to the Prescribing Information in Sri Lanka
Brief Title: Post-marketing Safety Study of GlaxoSmithKline (GSK) Biologicals' Synflorix™ Vaccine, in Healthy Infants and Children in Sri Lanka
Status: Withdrawn | Type: Observational
Why Stopped: Lack of clarity regarding the PMS study requirement from the RA and Ethics committee hence it was concluded GSK will submit local PSURs.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116290
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Immunisation Against Streptococcus Pneumoniae
Keywords: Post-marketing surveillance; Prescribing Information (PI); Healthy infants and children; Streptococcus pneumoniae; Synflorix™; Sri Lanka

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Synflorix™ cohort: Only those subjects to whom Synflorix™ will be administered as per normal clinical practice, according to the locally approved PI, will be included in the study.
  Interventions: Other: Synflorix™ data collection

INTERVENTIONS:
Other: Synflorix™ data collection — Safety monitoring and evaluation: recording of all AEs during the study period using diary cards, follow-up visit or telephone contact. Recording of SAEs throughout the study period for each subject.

SUMMARY:
This PMS study aims to collect safety and reactogenicity data of Synflorix™ in healthy infants and children of the local population as per the licensing requirement of the Sri Lankan regulatory authority.

DETAILED DESCRIPTION:
The participating physicians (investigators) will be asked to enrol only those subjects to whom they administer Synflorix™ in the course of their normal clinical practice according to the locally approved Prescribing Information.

Since there is lack of clarity regarding the PMS study requirement (both from Regulatory agency and Ethics Committee), it was decided that GSK will submit Local PSURs on a regular basis as desired by Local regulatory agency. The same is communicated to Regulatory agency and if they want something more they are requested to revert back with specific requirements.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/ LAR(s) can and will comply with the requirements of the protocol should be enrolled in the PMS study.
* Infants aged 6 weeks and above and children.
* Written, signed or thumb-printed informed consent obtained from the parent(s)/LAR(s) of the child. Where subject's parent(s)/LAR(s) are illiterate, the consent form will be countersigned by an impartial witness.

Note: Consent for this PMS study is solely for collection of safety and reactogenicity data and not for vaccination that is per routine practice. Data for demography, medical history and previous vaccination history, and concomitant medication/vaccination will also be collected.

Exclusion Criteria:

* Subjects with contraindications according to the locally approved PI.
* Child in care.
* Previous administration of three doses of Synflorix™.
* Previous vaccination with a pneumococcal vaccine other than Synflorix™.
* Planned administration of another pneumococcal vaccine other than Synflorix™ during the PMS study.

Ages: 6 Weeks to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy Sri Lankan infants aged 6 weeks and above and children
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of solicited local (any intensity) and general (any intensity and causally related) adverse events (AEs) | During the 4-day follow-up period (Day 0 to Day 3) following any dose of Synflorix™ and overall
Occurrence of unsolicited AEs | During the 31-day period (Day 0 to Day 30) following any dose of Synflorix™ and overall
Occurrence of Serious Adverse Events (SAEs) | Throughout the PMS study period, starting at Dose 1 (Visit 1) and ending 31 days (Day 0 to Day 30) after the last dose of Synflorix™ for each subject in the PMS study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline